CLINICAL TRIAL: NCT05309785
Title: Safety and Efficacy of Canagliflozin in Advanced CKD
Acronym: SIP-AKiD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Thomas Mavrakanas, Assistant Professor, Junior Scientist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-8410
Record Dates: First submitted 2022-03-14; First posted 2022-04-04 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: ESRD; CKD Stage 4; CKD Stage 5
Keywords: Canagliflozin; Advanced CKD; ESRD; Hemodialysis; Safety; Efficacy; SGLT-2 inhibitor
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — Canagliflozin; Tablets

STUDY DESIGN:
Intervention Model Description: We will conduct a single center, prospective, single-arm, open-label interventional study in 2 cohorts.
  Substudy 1: patients with advanced CKD, not yet on HD (N=36) Substudy 2: patients receiving HD (N=8)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Invokana 300 mg and 100 mg tablet — Substudy 1 Patients who fulfill the inclusion criteria and consent to participate will receive canagliflozin 100 mg po daily for 12+2 weeks (phase 1). For participants who have tolerated the drug, canagliflozin will be increased to 300 mg po daily for an additional 12+2 weeks (phase 2) and then stopped. If not tolerated, the dose will be reduced to 100 mg until the end of follow-up.
  Each phase of 12 weeks is followed by a 2-week window to ascertain surrogate efficacy outcomes.
  Substudy 2 Patients who fulfill the inclusion criteria and consent to participate will receive canagliflozin 100 mg po daily for 9 days.
  Other Names: Canagliflozin 300 mg and 100 mg tablet

SUMMARY:
The study objective is to characterize the pharmacokinetics (PK), pharmacodynamics, and surrogate measures of efficacy for canagliflozin in patients with advanced CKD, including those receiving HD.

As the CV and renoprotective effects of SGLT-2 inhibitors appear to be independent of glycemic control, the investigators hypothesize that canagliflozin will reduce albuminuria in patients with advanced CKD in the same manner as observed in patients with higher eGFR. The investigators also hypothesize that the 300 mg dose will be equally safe as the 100 mg dose but will have greater efficacy, given data which suggests efficacy correlates with drug exposure in patients without CKD.

Given its negligible renal elimination, the investigators hypothesize that exposure to canagliflozin 100 mg at steady state will not exceed the standard bioequivalence boundary of 80-125% in patients receiving HD, compared with published estimates with the 300 mg dose at steady state in individuals with preserved kidney function.

DETAILED DESCRIPTION:
Substudy 1:

Patients with eGFR<30 ml/min/1.73m2 and urine albumin to creatinine ratio (UACR)>200 mg/g not receiving dialysis will receive canagliflozin 100 mg po daily for 12 weeks (phase 1). For participants who have tolerated the drug, canagliflozin will be increased to 300 mg po daily for an additional 12 weeks (phase 2) and then stopped. Each phase will be followed by a 2-week window to ascertain surrogate efficacy outcomes.

Substudy 2:

Adult patients on HD for at least 3 months without significant residual renal function will receive canagliflozin 100 mg po daily for 9 days.

ELIGIBILITY:
Inclusion Criteria:

(Substudy 1- SIP-AKiD-1):

* adult patients with eGFR <30 ml/min/1.73m2
* urine albumin to creatinine ratio (UACR) >200 mg/g
* not receiving dialysis.

(Substudy 2- SIP-AKiD-2):

* adult patients on hemodialysis for at least 3 months
* without significant residual renal function, defined as a urine output <250 ml/24h.

Exclusion Criteria:

* Age <18 years
* type 1 diabetes
* history of euglycemic ketoacidosis
* known hypersensitivity to SGLT-2 inhibitors
* recurrent severe genital or urinary tract infections
* history of atraumatic amputation, gangrene, or active skin ulcer
* use within the last 48 h of an SGLT-2 inhibitor or a combined SGLT-1 and SGLT-2 inhibitor
* liver disease defined by an ALT > 3.0 times the upper limit of normal [ULN] or total bilirubin >1.5 times the ULN or liver cirrhosis of any stage
* gastrointestinal surgery or gastrointestinal disorder that could interfere with trial medication absorption
* pregnancy
* currently breastfeeding
* any other clinical condition that would jeopardize patient safety while participating in this trial.
* Patients receiving digoxin, phenobarbital, phenytoin, rifampin, or ritonavir will be excluded if these agents cannot be safely discontinued

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The 26-week change in albuminuria compared to baseline, as assessed by the UACR. | 26 weeks
  For substudy 1
The drug exposure at steady-state with 100 mg, as expressed by the AUC0-24, compared to published estimates with the 300 mg dose in patients with preserved renal function. | 8 days
  For substudy 2

SECONDARY OUTCOMES:
Change in UACR with 300 mg (at 26 weeks) vs. 100 mg dose (at 12 weeks) vs. baseline | At 12 and 26 weeks
  For substudy 1
Change in 24-hour ambulatory blood pressure (BP) | At 12 and 26 weeks
  For substudy 1
Area under the plasma concentration versus time curve (AUC) | At 12 and 26 weeks
  For substudy 1
Change in 6-minute walk distance from baseline | At 12 and 26 weeks
  For substudy 1
Change in urinary excretion of sodium from baseline | At 12 and 26 weeks
  For substudy 1
Neutrophil gelatinase-associated lipocalin (NGAL) levels | After ≥12 weeks of treatment with each dose
  For substudy 1

OTHER OUTCOMES:
Change in urinary excretion of phosphate from baseline | After ≥12 weeks of treatment with each dose
  For substudy 1
Peak plasma concentration (Cmax) | 8 days
  For substudy 2
Time to peak plasma concentration (tmax) | 8 days
  For substudy 2
Trough plasma concentration (Cmin) | 8 days
  For substudy 2
Effective half-life (t1/2) | 8 days
  For substudy 2

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Mavrakanas, MD, Principal Investigator — Research Institute of the McGill University Health Center
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Elenjickal EJ, Mavrakanas TA, Gritsas A, Suri RS, Marsot A. Population Pharmacokinetic Modeling of Canagliflozin in Advanced Chronic Kidney Disease. Clin Pharmacokinet. 2025 Nov;64(11):1693-1708. doi: 10.1007/s40262-025-01571-8. Epub 2025 Sep 15. PMID 40952584